CLINICAL TRIAL: NCT01562314
Title: A Randomised, Double-blind, Placebo-controlled Parallel Group, Pilot Study of GWP42003 in the Symptomatic Treatment of Ulcerative Colitis
Brief Title: A Pilot Study of GWP42003 in the Symptomatic Treatment of Ulcerative Colitis (GWID10160)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GW Research Ltd (Industry)
Responsible Party: Sponsor
Organization: GWResearch (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GWID10160; 2011-003208-19 (EudraCT Number)
Record Dates: First submitted 2012-03-21; First posted 2012-03-23 (Estimated); Results first posted 2015-08-14 (Estimated); Last update posted 2018-08-09 (Actual); Status verified 2018-07

CONDITIONS: Ulcerative Colitis
Keywords: Mild to Moderate Ulcerative Colitis; GWP42003
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- GWP42003 (Experimental): GWP42003 was administered orally at a dose of 50 mg up to 250 mg, BID, in the fasted state in the morning and evening, for 10 weeks. Following randomization, participants entered a 2-week dose escalation period to achieve their maximum tolerated dose, up to 500 mg, and maintained this dose for the rest of the treatment period. Participants were then followed for 1 week.
  Interventions: Drug: GWP42003
- Placebo (Placebo Comparator): Placebo capsules matching the study drug were administered orally, BID, in the fasted state in the morning and evening, for 10 weeks. Participants were then followed for 1 week.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GWP42003 — 1 to 5 50 mg capsules taken BID
  Other Names: Cannabidiol (CBD) Botanical Drug Substance (BDS)
  Arms: GWP42003
Drug: Placebo — 1 to 5 matching capsules taken BID
  Other Names: Placebo control
  Arms: Placebo

SUMMARY:
This study was conducted to determine the efficacy and safety of GWP42003 compared with placebo by the percentage of participants achieving remission quantified as a Mayo score of 2 or less (with no sub-score >1) after 10 weeks of treatment.

DETAILED DESCRIPTION:
This study was conducted by GW Research Ltd as a pilot study to determine the efficacy and safety of GWP42003 (50 milligram [mg] up to 250 mg twice daily [BID]), compared with placebo, as assessed by the percentage of participants achieving remission quantified as a Mayo score of 2 or less (with no sub-score >1) after 10 weeks of treatment. This was the first study to determine whether the study drug has a positive benefit for participants on their ulcerative colitis symptom control, as well as effects on inflammatory marker cytokines (C reactive protein [CRP]), a fecal inflammatory marker (calprotectin), stool frequency, and rectal bleeding. In addition, various inflammatory bowel disease (IBD) questionnaires were implemented in the study to observe further benefits on the study drug, compared with placebo.

This study was multi-center, randomized, double-blind, placebo-controlled, and parallel-group. The study consisted of a 7-day baseline period, a 10-week treatment period, and a 1-week follow-up period. Each participant had a Mayo assessment (including endoscopy) conducted to confirm eligibility. Eligible participants were randomized in a 1:1 ratio into the GWP42003 and placebo groups. At the start of the treatment period, participants entered a 2-week dose escalation period to achieve their maximum tolerated dose, up to 250 mg BID in the GWP42003 group. Participants remained at the maximum tolerated dose for the rest of the treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants aged 18 years or above;
* Participant diagnosed with mild to moderate ulcerative colitis and on a fixed dose of 5-Aminosalicylic (5-ASA) treatment and have been on a stable dose for at least 2 weeks prior to screening (0 mg dose of 5-ASA was acceptable);
* Participants at screening and baseline with a Mayo assessment score of greater than or equal to 4 (≥4) but less than or equal to 10 (≤10) and with an endoscopy score of at least 1 (≥1) , following an adequate exposure to oral and/ or topical 5-ASA, in the opinion of the investigator;
* In the opinion of the investigator, capable of complying with the study requirements and completing the study;
* Willing and able to give informed consent;
* Willing for his or her name to be notified to the responsible authorities for participation in this study, as applicable;
* Willing to allow his or her primary care practitioner and consultant, if appropriate, to be notified of participation in the study;

Exclusion Criteria:

* Severe ulcerative colitis (Mayo score of greater than 10 (>10);
* Ulcerative colitis only affecting the rectum (proctitis)
* Gastrointestinal infection evident from stool culture and testing for Clostridium difficile toxin (in the opinion of the investigator);
* Currently using or had used recreational cannabis, medicinal cannabis, cannabinoid medications (including Sativex®), or synthetic cannabinoid-based medications within 1 month prior to study entry and unwilling to abstain for the duration of the study;
* Any known or suspected history of alcohol or substance abuse, epilepsy or recurrent seizures, or hypersensitivity to cannabinoids;
* Was receiving a prohibited medication prior to screening and for the duration of the study;
* Previous non-responders to mono or polyclonal anti-Tumor Necrosis Factor antibodies;
* Personal or first degree relative, with history of schizophrenia or other psychosis;
* History of other significant psychiatric disorder or severe personality disorder (at the discretion of the investigator);
* Any known or suspected history of depression sufficient to require treatment with antidepressants or disrupt ordinary life (excluding episodes of reactive depression at the discretion of the investigator);
* Clinically significant cardiac, renal or hepatic impairment in the opinion of the investigator;
* Female participants who were pregnant, lactating or planning pregnancy during the course of the study and for 3 months from the date of last dose;
* Female participants of child bearing potential, unless willing to use 2 forms of contraception, 1 of which must have been a barrier contraception (for example, a female condom or occlusive cap [diaphragm or cervical vault/caps] with spermicide) during the study and for 3 months from the date of last dose (however a male condom should not have been used in conjunction with the female condom);
* Male participants whose partner was of child bearing potential, unless willing to use an appropriate barrier method of contraception (condom and spermicide) in addition to having their female partner use another form of barrier contraception (for example, an occlusive cap [diaphragm or cervical vault/caps] with spermicide) during the study and for 3 months from date of last dose (however a male condom should not have been used in conjunction with a female condom);
* Planned to travel outside the country of residence during the treatment phase of the study;
* Received an Investigational Medicinal Product (IMP) within 30 days prior to the screening visit;
* In the opinion of the investigator, was not considered to be suitable for the study;
* Any other significant disease or disorder which, in the opinion of the investigator, may either have put the participant at risk because of participation in the study, or may have influenced the result of the study or the participant's ability to participate in the study;
* Participant with any abnormalities that, in the opinion of the investigator, would prevent the participant from safe participation in the study;
* Unwilling to abstain from donation of blood during the study;
* Participants previously randomized into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-05-09 (Actual); Primary Completion 2014-08-05 (Actual); Study Completion 2014-08-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United Kingdom (6):
  - Birmingham
  - Coventry
  - Liverpool
  - London
  - Middlesex
  - Wigan

REFERENCES:
- [Result] Irving PM, Iqbal T, Nwokolo C, Subramanian S, Bloom S, Prasad N, Hart A, Murray C, Lindsay JO, Taylor A, Barron R, Wright S. A Randomized, Double-blind, Placebo-controlled, Parallel-group, Pilot Study of Cannabidiol-rich Botanical Extract in the Symptomatic Treatment of Ulcerative Colitis. Inflamm Bowel Dis. 2018 Mar 19;24(4):714-724. doi: 10.1093/ibd/izy002. PMID 29538683

RESULTS

PARTICIPANT FLOW:
Groups:
- GWP42003: GWP42003 was administered orally at a dose of 50 milligram (mg) up to 250 mg, twice daily (BID), in the fasted state in the morning and evening, for 10 weeks. Following randomization, participants entered a 2-week dose escalation period to achieve their maximum tolerated dose, up to 500 mg, and maintained this dose for the rest of the treatment period. Participants were then followed for 1 week.
Period: Overall Study
Arm/Group | GWP42003 | Placebo
Started | 29 | 31
Received at Least 1 Dose of Study Drug (Safety analysis set; participants analyzed according to treatment received.) | 29 | 31
Intent-to-Treat (ITT) Analysis Set (All randomized participants who received ≥1 dose of study drug; analyzed by randomization group.) | 29 | 31
Per Protocol (PP) Analysis Set (All participants without protocol violations that compromised the assessments of efficacy.) | 17 | 27
Completed | 16 | 23
Not Completed | 13 | 8
Not completed — Adverse Event | 10 | 5
Not completed — Met Withdrawal Criteria | 3 | 2
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) analysis set: all participants who were randomized and received at least 1 dose of study drug. Participants were analyzed according to the group to which they were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | GWP42003 | Placebo | Total
Number analyzed (Participants) | 29 | 31 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.78 (15.050) | 42.82 (12.916) | 43.77 (13.903)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 10 | 16
  Male | 23 | 21 | 44

OUTCOME MEASURES:

1. Primary Outcome: Number Of Participants With A Mayo Score Of 2 Or Less (With No Sub-score >1) At EOT
Description: The Mayo score is an assessment of ulcerative colitis activity. The Mayo total score ranges from 0 to 12 points with higher scores indicating more severe disease. The total score is made up of 4 sub-scores, each of which is assessed using a 0 to 3 scale. Sub-scores are graded as follows: Stool Frequency: 0 = Normal number of stools, 1 = 1 to 2 stools more than normal, 2 = 3 to 4 stools more than normal, 3 = 5 or more stools more than normal; Rectal Bleeding: 0 = No blood seen, 1 = Streaks of blood with stool less than half the time, 2 = Obvious blood with stool most of the time or more, 3 = Blood alone passes; Findings on Endoscopy: 0 = Normal or inactive disease, 1 = Mild disease (erythema, decreased vascular pattern, mild friability), 2 = Moderate disease (marked erythema, lack of vascular pattern, friability, erosions), 3 = Severe disease (spontaneous bleeding, ulceration); Physician's Global Assessment of Illness Severity (PGAS): 0 = none, 1 = mild, 2 = moderate, and 3 = severe.
Time Frame: Baseline to End of Treatment (EOT) (10 weeks) or Early Termination (ET)
Population: ITT analysis set: all participants who were randomized and received at least 1 dose of study drug. Participants were analyzed according to the group to which they were randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | GWP42003 | Placebo
Number analyzed (Participants) | 29 | 31
Participants | 8 | 8
Statistical Analysis 1: Comparison: GWP42003 vs Placebo; Test type: Superiority or Other; p = 0.7532, Regression, Logistic; Odds Ratio (OR) = 0.821, 90% CI 2-sided [0.292 to 2.309]

2. Primary Outcome: Number Of Participants With A Mayo Score Of 2 Or Less (With No Sub-score >1) At EOT - PP Analysis
Description: The Mayo score is an assessment of ulcerative colitis activity. The Mayo total score ranges from 0 to 12 points with higher scores indicating more severe disease. The total score is made up of 4 sub-scores, each of which is assessed using a 0 to 3 scale. Sub-scores are graded as follows: Stool Frequency: 0 = Normal number of stools, 1 = 1 to 2 stools more than normal, 2 = 3 to 4 stools more than normal, 3 = 5 or more stools more than normal; Rectal Bleeding: 0 = No blood seen, 1 = Streaks of blood with stool less than half the time, 2 = Obvious blood with stool most of the time or more, 3 = Blood alone passes; Findings on Endoscopy: 0 = Normal or inactive disease, 1 = Mild disease (erythema, decreased vascular pattern, mild friability), 2 = Moderate disease (marked erythema, lack of vascular pattern, friability, erosions), 3 = Severe disease (spontaneous bleeding, ulceration); PGAS: 0 = none, 1 = mild, 2 = moderate, and 3 = severe.
Time Frame: Baseline to EOT (10 weeks) or ET
Population: PP analysis set: all participants who completed the 10-week randomized phase of the study with no protocol violations deemed to compromise the assessments of efficacy.
Measure: Count of Participants; unit: Participants
Arm/Group | GWP42003 | Placebo
Number analyzed (Participants) | 17 | 27
Participants | 7 | 8
Statistical Analysis 1: Comparison: GWP42003 vs Placebo; Test type: Superiority or Other; p = 0.7032, Regression, Logistic; Odds Ratio (OR) = 1.300, 90% CI 2-sided [0.419 to 4.040]

3. Secondary Outcome: Distribution On The PGAS At EOT
Description: The PGAS required the physician to assess participants' disease severity on a 4-point scale (0=normal [no disease], 1 = mild disease, 2 = moderate disease, 3 = severe disease).
Time Frame: EOT (10 weeks) or ET
Population: ITT analysis set: all participants who were randomized and received at least 1 dose of study drug. Participants were analyzed according to the group to which they were randomized. Not all participants contributed data for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | GWP42003 | Placebo
Number analyzed (Participants) | 26 | 31
Participants
  Normal | 7 | 5
  Mild Disease | 13 | 11
  Moderate Disease | 6 | 12
  Severe Disease | 0 | 3

4. Secondary Outcome: Distribution On The PGAS At EOT - PP Analysis
Description: The PGAS required the physician to assess participants' disease severity on a 4-point scale (0 = normal [no disease], 1 = mild disease, 2 = moderate disease, 3 = severe disease).
Time Frame: EOT (10 weeks) or ET
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GWP42003 | Placebo
Number analyzed (Participants) | 17 | 27
Participants
  Normal | 6 | 5
  Mild Disease | 8 | 9
  Moderate Disease | 3 | 11
  Severe Disease | 0 | 2

5. Secondary Outcome: Change From Baseline To EOT In The PGAS Score
Description: The PGAS required the physician to assess participants' disease severity on a 4-point scale (0=normal [no disease], 1 = mild disease, 2 = moderate disease, 3 = severe disease). A negative change from Baseline indicates that symptoms decreased.
Time Frame: Baseline to EOT (10 weeks) or ET
Population: ITT analysis set: all participants who were randomized and received at least 1 dose of study drug. Participants were analyzed according to the group to which they were randomized. Not all participants contributed data to this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GWP42003 | Placebo
Number analyzed (Participants) | 29 | 31
units on a scale
  Baseline | 1.7 (0.45) | 1.8 (0.48)
  Final Visit: number analyzed (Participants) | 26 | 31
  Final Visit | 1.0 (0.72) | 1.4 (0.89)
  Change From Baseline: number analyzed (Participants) | 26 | 31
  Change From Baseline | -0.8 (0.82) | -0.4 (0.95)

6. Secondary Outcome: Change From Baseline To EOT In The PGAS Score - PP Analysis
Description: as for outcome 5
Time Frame: Baseline to EOT (10 weeks) or ET
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GWP42003 | Placebo
Number analyzed (Participants) | 17 | 27
units on a scale
  Baseline | 1.8 (0.44) | 1.8 (0.51)
  Final Visit | 0.8 (0.73) | 1.4 (0.88)
  Change From Baseline | -0.9 (0.83) | -0.4 (0.97)

7. Secondary Outcome: Change From Baseline To EOT In The Inflammatory Bowel Disease Questionnaire (IBDQ) Total Score
Description: The IBDQ is a validated and reliable tool to measure health-related quality of life in adult participants with inflammatory bowel disease (IBD). Each of the 32 questions falls into 1 of 4 domains (bowel symptoms, systemic symptoms, emotional status and social function). The 32 questions each have 7 possible responses. Each response is assigned a score ranging from 1 to 7, indicating the severity (1 being least favorable and 7 being the most favorable). Individual question scores were summed to give the IBDQ total score (range: 32 to 224 points). A positive change from Baseline indicates that symptoms improved.
Time Frame: Baseline to EOT (10 weeks) or ET
Population: ITT analysis set: all participants who were randomized and received at least 1 dose of study drug. Participants were analyzed according to the group to which they were randomized. Not all participants contributed data for the outcome measure.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | GWP42003 | Placebo
Number analyzed (Participants) | 29 | 31
units on a scale
  Baseline: number analyzed (Participants) | 24 | 30
  Baseline | 138.5 (32.37) | 129.1 (38.02)
  Final Visit: number analyzed (Participants) | 29 | 30
  Final Visit | 164.2 (29.13) | 146.8 (47.50)
  Change From Baseline: number analyzed (Participants) | 24 | 29
  Change From Baseline | 24.6 (35.51) | 16.7 (36.33)

8. Secondary Outcome: Change From Baseline To EOT In The IBDQ Total Score - PP Analysis
Description: The IBDQ is a validated and reliable tool to measure health-related quality of life in adult participants with IBD. Each of the 32 questions falls into 1 of 4 domains (bowel symptoms, systemic symptoms, emotional status and social function). The 32 questions each have 7 possible responses. Each response is assigned a score ranging from 1 to 7, indicating the severity (1 being least favorable and 7 being the most favorable). Individual question scores were summed to give the IBDQ total score (range: 32 to 224 points). A positive change from Baseline indicates that symptoms improved.
Time Frame: Baseline to EOT (10 weeks) or ET
Population: PP analysis set: all participants who completed the 10-week randomized phase of the study with no protocol violations deemed to compromise the assessments of efficacy. Not all participants contributed data for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GWP42003 | Placebo
Number analyzed (Participants) | 17 | 27
units on a scale
  Baseline: number analyzed (Participants) | 14 | 26
  Baseline | 134.0 (35.58) | 134.0 (37.30)
  Final Visit: number analyzed (Participants) | 17 | 26
  Final Visit | 172.8 (28.52) | 150.5 (48.87)
  Change From Baseline: number analyzed (Participants) | 14 | 25
  Change From Baseline | 39.3 (39.81) | 15.4 (33.65)

9. Secondary Outcome: Number Of Participants Who Reported An Improvement In The Subject Global Impression Of Change (SGIC) Questionnaire At EOT
Description: Participants were asked to answer the following question by using a 7-point scale (1 = very much better to 7 = very much worse): "Please assess the change in your ulcerative colitis symptoms since immediately before receiving the first dose of study treatment." Improvement was considered as very much better, much better, or minimally better.
Time Frame: Visit 4 (Day 43) to EOT (10 weeks) or ET
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | GWP42003 | Placebo
Number analyzed (Participants) | 29 | 31
Participants
  Visit 4 (Day 43): number analyzed (Participants) | 18 | 25
  Visit 4 (Day 43) | 15 | 18
  Final Visit | 23 | 17

10. Secondary Outcome: Number Of Participants Who Reported An Improvement In The SGIC Questionnaire At EOT - PP Analysis
Description: as for outcome 9
Time Frame: Visit 4 (Day 43) to EOT (10 weeks) or ET
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | GWP42003 | Placebo
Number analyzed (Participants) | 17 | 27
Participants
  Visit 4 (Day 43): number analyzed (Participants) | 17 | 25
  Visit 4 (Day 43) | 14 | 18
  Final Visit | 16 | 16

11. Secondary Outcome: Change From Baseline To The Last Week Of Treatment In Ulcerative Colitis Symptoms, As Measured By Scores On The Stool Frequency Numerical Rating Scale (NRS)
Description: Participants were required to record their stool frequency during the baseline and treatment periods in a daily diary. Participants graded stool frequency with a 4-point NRS as follows: 0 = Normal number of stools; 1 = 1 to 2 stools more than normal; 2 = 3 to 4 stools more than normal; 3 = 5 or more stools more than normal. For analysis, the baseline value was defined as the mean stool frequency score of the last 7 available days of the baseline period; the EOT value was defined as the mean stool frequency score of last 7 days of the treatment period, or last 7 days for which study drug was taken, where earlier. A negative change from Baseline indicates that symptoms improved.
Time Frame: Baseline to EOT (last 7 days) or ET
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GWP42003 | Placebo
Number analyzed (Participants) | 29 | 31
units on a scale
  Baseline | 1.50 (0.937) | 1.89 (0.814)
  Last 7 Days: number analyzed (Participants) | 28 | 31
  Last 7 Days | 1.05 (0.930) | 1.46 (0.888)
  Change From Baseline: number analyzed (Participants) | 28 | 31
  Change From Baseline | -0.43 (0.563) | -0.43 (0.816)

12. Secondary Outcome: Change From Baseline To The Last Week Of Treatment In Ulcerative Colitis Symptoms, As Measured By Scores On The Stool Frequency NRS - PP Analysis
Description: as for outcome 11
Time Frame: Baseline to EOT (last 7 days) or ET
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GWP42003 | Placebo
Number analyzed (Participants) | 17 | 27
units on a scale
  Baseline | 1.37 (0.875) | 1.81 (0.827)
  Last 7 Days | 0.73 (0.689) | 1.36 (0.871)
  Change From Baseline | -0.64 (0.497) | -0.45 (0.768)

13. Secondary Outcome: Change From Baseline To The Last Week Of Treatment In Ulcerative Colitis Symptoms, As Measured By Scores On The Rectal Bleeding NRS
Description: Participants were required to record their rectal bleeding during the baseline and treatment periods in a daily diary. Participants graded rectal bleeding with a 4-point NRS as follows: 0 = No blood seen, 1 = Streaks of blood with stool less than half the time, 2 = Obvious blood with stool most of the time or more, 3 = Blood alone passes. For analysis, the baseline value was defined as the mean rectal bleeding score of the last 7 available days of the baseline period; the EOT value was defined as the mean rectal bleeding score of last 7 days of the treatment period, or last 7 days for which study drug was taken, where earlier. A negative change from Baseline indicates that symptoms improved.
Time Frame: Baseline to EOT (last 7 days) or ET
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GWP42003 | Placebo
Number analyzed (Participants) | 29 | 31
units on a scale
  Baseline | 0.96 (0.829) | 1.19 (0.816)
  Last 7 Days: number analyzed (Participants) | 28 | 31
  Last 7 Days | 0.48 (0.711) | 0.84 (0.863)
  Change From Baseline: number analyzed (Participants) | 28 | 31
  Change From Baseline | -0.44 (0.709) | -0.35 (0.794)

14. Secondary Outcome: Change From Baseline To The Last Week Of Treatment In Ulcerative Colitis Symptoms, As Measured By Scores On The Rectal Bleeding NRS - PP Analysis
Description: as for outcome 13
Time Frame: Baseline to EOT (last 7 days) or ET
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GWP42003 | Placebo
Number analyzed (Participants) | 17 | 27
units on a scale
  Baseline | 0.82 (0.682) | 1.16 (0.831)
  Last 7 Days | 0.24 (0.367) | 0.80 (0.875)
  Change From Baseline | -0.58 (0.793) | -0.35 (0.773)

15. Secondary Outcome: Change From Baseline To EOT In The Mayo Total Score
Description: The Mayo score is an assessment of ulcerative colitis activity. The Mayo total score ranges from 0 to 12 points with higher scores indicating more severe disease. The total score is made up of 4 sub-scores (assessed using a 0 to 3 scale). The sub-scores are graded as follows: Stool Frequency: 0 = Normal number of stools, 1 = 1 to 2 stools more than normal, 2 = 3 to 4 stools more than normal, 3 = 5 or more stools more than normal; Rectal Bleeding: 0 = No blood seen, 1 = Streaks of blood with stool less than half the time, 2 = Obvious blood with stool most of the time or more, 3 = Blood alone passes; Findings on Endoscopy: 0 = Normal or inactive disease, 1 = Mild disease (erythema, decreased vascular pattern, mild friability), 2 = Moderate disease (marked erythema, lack of vascular pattern, friability, erosions), 3 = Severe disease (spontaneous bleeding, ulceration); PGAS: 0 = none, 1 = mild, 2 = moderate and 3 = severe. A negative change from Baseline indicates that symptoms improved.
Time Frame: Baseline to EOT (10 weeks) or ET
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GWP42003 | Placebo
Number analyzed (Participants) | 29 | 31
units on a scale
  Baseline | 6.3 (1.73) | 7.0 (2.01)
  Final Visit: number analyzed (Participants) | 21 | 26
  Final Visit | 3.0 (2.25) | 4.9 (3.22)
  Change From Baseline: number analyzed (Participants) | 21 | 26
  Change From Baseline | -3.0 (2.40) | -1.8 (2.73)

16. Secondary Outcome: Change From Baseline To EOT In The Mayo Partial Score
Description: The Mayo score is an assessment of ulcerative colitis activity. The Mayo partial score does not include the endoscopy findings sub-score and ranges from 0 to 9 points with higher scores indicating more severe disease. The partial score is made up of 3 sub-scores (assessed by using a 0 to 3 scale). The sub-scores are graded as follows: Stool Frequency: 0 = Normal number of stools, 1 = 1 to 2 stools more than normal, 2 = 3 to 4 stools more than normal, 3 = 5 or more stools more than normal; Rectal Bleeding: 0 = No blood seen, 1 = Streaks of blood with stool less than half the time, 2 = Obvious blood with stool most of the time or more, 3 = Blood alone passes; PGAS: 0 = none, 1 = mild, 2 = moderate and 3 = severe. A negative change from Baseline indicates that symptoms improved.
Time Frame: Baseline to EOT (10 weeks) or ET
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GWP42003 | Placebo
Number analyzed (Participants) | 29 | 31
units on a scale
  Baseline | 4.4 (1.57) | 5.1 (1.61)
  Final Visit: number analyzed (Participants) | 26 | 30
  Final Visit | 2.3 (1.73) | 3.8 (2.60)
  Change From Baseline: number analyzed (Participants) | 26 | 30
  Change From Baseline | -2.0 (2.00) | -1.2 (2.14)

17. Secondary Outcome: Change From Baseline To EOT In Levels Of Fecal Calprotectin
Description: Fecal calprotectin is a marker of inflammation. Standard methods were used to measure the levels of calprotectin in fecal samples collected at the end of baseline and treatment periods. A negative change from Baseline indicates that levels of fecal calprotectin decreased.
Time Frame: Baseline to EOT (10 weeks) or ET
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: microgram calprotectin/gram feces (ug/g)
Arm/Group | GWP42003 | Placebo
Number analyzed (Participants) | 29 | 31
microgram calprotectin/gram feces (ug/g)
  Baseline: number analyzed (Participants) | 27 | 29
  Baseline | 490.6 (197.41) | 462.3 (227.35)
  Final Visit: number analyzed (Participants) | 23 | 30
  Final Visit | 397.3 (241.08) | 428.0 (229.38)
  Change from Baseline: number analyzed (Participants) | 22 | 28
  Change from Baseline | -91.6 (295.77) | -51.3 (289.32)

18. Post Hoc Outcome: Change From Baseline To EOT In The Mayo Total Score - PP Analysis
Description: The Mayo score is an assessment of ulcerative colitis activity. The Mayo total score ranges from 0 to 12 points with higher scores indicating more severe disease. The total score is made up of 4 sub-scores (assessed using a 0 to 3 scale). The sub-scores are graded as follows: Stool Frequency: 0 = Normal number of stools, 1 = 1 to 2 stools more than normal, 2 = 3 to 4 stools more than normal, 3 = 5 or more stools more than normal; Rectal Bleeding: 0 = No blood seen, 1 = Streaks of blood with stool less than half the time, 2 = Obvious blood with stool most of the time or more, 3 = Blood alone passes; Findings on Endoscopy: 0 = Normal or inactive disease, 1 = Mild disease (erythema, decreased vascular pattern, mild friability), 2 = Moderate disease (marked erythema, lack of vascular pattern, friability, erosions), 3 = Severe disease (spontaneous bleeding, ulceration); PGAS: 0 = none, 1 = mild, 2 = moderate, and 3 = severe. A negative change from Baseline indicates that symptoms improved.
Time Frame: Baseline to EOT (10 weeks) or ET
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GWP42003 | Placebo
Number analyzed (Participants) | 17 | 27
units on a scale
  Baseline | 6.0 (1.70) | 6.8 (2.04)
  Final Visit: number analyzed (Participants) | 17 | 24
  Final Visit | 2.8 (2.02) | 4.7 (3.24)
  Change From Baseline: number analyzed (Participants) | 17 | 24
  Change From Baseline | -3.2 (2.25) | -1.9 (2.81)

19. Post Hoc Outcome: Change From Baseline To EOT In The Mayo Partial Score - PP Analysis Set
Description: The Mayo score is an assessment of ulcerative colitis activity. The Mayo partial score does not include the endoscopy findings sub-score and ranges from 0 to 9 points with higher scores indicating more severe disease. The partial score is made up of 3 sub-scores (assessed by using a 0 to 3 scale). The sub-scores are graded as follows: Stool Frequency: 0 = Normal number of stools, 1 = 1 to 2 stools more than normal, 2 = 3 to 4 stools more than normal, 3 = 5 or more stools more than normal; Rectal Bleeding: 0 = No blood seen, 1 = Streaks of blood with stool less than half the time, 2 = Obvious blood with stool most of the time or more, 3 = Blood alone passes; PGAS: 0 = none, 1 = mild, 2 = moderate, and 3 = severe. A negative change from Baseline indicates that symptoms improved.
Time Frame: Baseline to EOT (10 weeks) or ET
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GWP42003 | Placebo
Number analyzed (Participants) | 17 | 27
units on a scale
  Baseline | 4.1 (1.50) | 4.9 (1.63)
  Final Visit | 1.7 (1.53) | 3.7 (2.66)
  Change From Baseline | -2.4 (2.03) | -1.2 (2.17)

20. Post Hoc Outcome: Change From Baseline To EOT In Levels Of Fecal Calprotectin- PP Analysis
Description: as for outcome 17
Time Frame: Baseline to EOT (10 weeks) or ET
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: ug/g
Arm/Group | GWP42003 | Placebo
Number analyzed (Participants) | 17 | 27
ug/g
  Baseline: number analyzed (Participants) | 16 | 25
  Baseline | 527.9 (164.14) | 440.3 (237.99)
  Final Visit: number analyzed (Participants) | 17 | 26
  Final Visit | 355.9 (247.75) | 408.9 (238.94)
  Change From Baseline: number analyzed (Participants) | 16 | 24
  Change From Baseline | -155.9 (306.84) | -51.9 (311.56)

ADVERSE EVENTS:
Time Frame: Post-dose on Day 1 through 14 days after the final dose (up to 85 days).
Description: Safety analysis set: All randomized participants who received at least one dose of study drug and were analyzed according to the treatment received.
Arm/Group | GWP42003 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/29 | 4/31
Other Adverse Events (participants affected / at risk) | 28/29 | 23/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | GWP42003 (N=29) | Placebo (N=31)
Colitis ulcerative (Gastrointestinal disorders) | 0 | 2
Chest pain (General disorders) | 0 | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0/6 | 1/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GWP42003 (N=29) | Placebo (N=31)
Palpitations (Cardiac disorders) | 2 | 0
Abdominal discomfort (Gastrointestinal disorders) | 2 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 3
Abdominal pain (Gastrointestinal disorders) | 1 | 5
Colitis (Gastrointestinal disorders) | 1 | 3
Colitis ulcerative (Gastrointestinal disorders) | 1 | 3
Constipation (Gastrointestinal disorders) | 0 | 3
Dry mouth (Gastrointestinal disorders) | 4 | 0
Nausea (Gastrointestinal disorders) | 8 | 3
Vomiting (Gastrointestinal disorders) | 4 | 0
Fatigue (General disorders) | 4 | 4
Lower respiratory tract infection (Infections and infestations) | 3 | 0
Nasopharyngitis (Infections and infestations) | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Muscle twitching (Musculoskeletal and connective tissue disorders) | 2 | 0
Disturbance in attention (Nervous system disorders) | 5 | 0
Dizziness (Nervous system disorders) | 12 | 3
Headache (Nervous system disorders) | 4 | 4
Lethargy (Nervous system disorders) | 2 | 2
Memory impairment (Nervous system disorders) | 3 | 0
Somnolence (Nervous system disorders) | 10 | 2
Disorientation (Psychiatric disorders) | 4 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 180 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.